CLINICAL TRIAL: NCT00793741
Title: Measurement of Glucose Metabolism in Humans Using Magnetic Resonance at 4 Tesla. Substudy: Hypoglycemia Unawareness
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 9711M00055
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Type 1 Diabetes; Hypoglycemia Unawareness
Keywords: Type 1 diabetes; Hypoglycemia unawareness; Islet transplant
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Somatostatin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Type 1 Diabetes Hypoglycemia unawareness Islet transplant candidate
  Interventions: Drug: somatostatin
- 2: Healthy control subjects
  Interventions: Drug: somatostatin

INTERVENTIONS:
Drug: somatostatin — Somatostatin may be used to suppress endogenous insulin secretion

SUMMARY:
The purpose of this study is to determine whether islet transplantation alters brain glucose concentrations in patients with type 1 diabetes, recurrent hypoglycemia, and hypoglycemia unawareness when compared to that measured prior to transplant in the same subjects.

DETAILED DESCRIPTION:
Individuals with type 1 diabetes and hypoglycemia unawareness who become active islet transplant candidates and matched controls will be recruited for participation in this study. Subjects will undergo a hyperglycemic clamp with somatostatin before and 6 months after islet transplantation. During the clamp study, their brain glucose concentrations will be measured by proton magnetic resonance spectroscopy. Following these measurements, subjects will undergo a hypoglycemic clamp study to assess their counterregulatory response.

On the morning of the study subjects will report to the Clinical Research Center in the CMRR and be asked to do the following:

1. All subjects will be asked not to eat anything after midnight on the day before the magnet study at the Magnet Center. A small plastic catheter will be placed in a vein in each arm for infusion of hormones. A third plastic catheter will be placed in a foot vein for measuring blood glucose levels. The foot and distal leg will be placed in a heated blanket for the duration of the study to speed up the flow of blood through the vein and for easy withdrawing of blood. During the study subjects will receive carefully calculated doses of insulin, glucose, potassium phosphate, and somatostatin. These substances will be contained in syringes or bags and pumped through intravenous catheters placed in the arms. Insulin and somatostatin are hormones that are made naturally by the body. Initially we will keep blood sugar at the normal level. The blood glucose will then be raised by infusing glucose at a calculated rate. We will maintain the high blood sugar concentration for 45 to 120 minutes. This causes no symptoms other than a necessity f to pass urine more frequently than normal. The blood glucose infusion will then be dropped to allow blood glucose to drop in small steps to the normal glucose concentration. We will draw at most 15 oz. of blood during this part of the study.
2. All subjects will be asked to participate in a second experiment after the magnet study. Subjects may chose to perform this part of the study at Yale University. If subjects choose to stay at the University Of Minnesota, they will be participating in the second experiment either the same day or the day after the first experiment. If done the same day, the arm catheters will be left in place for infusion of insulin, potassium phosphate, and glucose. A third catheter may be placed in the hand for venous blood sampling. This hand will be placed in a warming box to ensure adequate blood flow and accurate laboratory results. Blood will be drawn every 5 minutes for measurement of glucose and other hormones. The total amount of blood drawn will be about 10 tablespoons. Insulin will be infused to lower blood sugar level to a level below the normal range. It will be maintained at this low level for thirty minutes after which time the insulin infusion will be discontinued and the blood sugar level allowed to normalize. Subjects will then be given a meal.
3. Subjects with type 1 diabetes will be asked to spend the night before each study at the General Clinical Research Center so that blood glucose values can be maintained between 80-110 mg/dl. They will be asked to hold insulin doses in the evening before and on the morning of the study and insulin will be provided via an intravenous infusion. For those subjects with diabetes who chose to undergo all testing at the University of Minnesota, they will be followed as inpatients in the GCRC during one to two days of testing.
4. Following islet transplant subjects will be asked to undergo the magnet study described under point #1 above and the hypoglycemia study described under point #3 above at approximately 3-9 months after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Must be able to provide informed consent
* Type 1 diabetes >5 years duration
* Healthy controls

Exclusion Criteria:

* Over 300 pounds
* Claustrophobic
* History of ischemic heart disease, arrhythmia or seizure disorder
* Pregnant
* On medications known to alter blood flow or carbohydrate metabolism
* Have internally located pieces of metal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Endocrinology clinic, community
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Brain glucose concentration as measured by NMR spectroscopy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States